CLINICAL TRIAL: NCT05512312
Title: Treatment of Excessive Gingival Display Using Conventional Esthetic Crown Lengthening Versus Computer Guided Esthetic Crown Lengthening: (A Randomized Clinical Trial)
Brief Title: Computer Guided Esthetic Crown Lengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Borham, Teaching Assistant, Faculty of Dentistry, Misr International University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Guided gummy smile correction
Record Dates: First submitted 2022-06-05; First posted 2022-08-23 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2022-12

CONDITIONS: Altered Passive Eruption of Teeth; Guided Surgery; Gummy Smile

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Eight patients indicated for ECL were treated using digitally assisted crown lengthening utilizing 3D printed surgical stents.
  Interventions: Procedure: Computer guided Esthetic crown lengthening
- Control Group (Active Comparator): Eight patients indicated for ECL were managed by conventional crown lengthening.
  Interventions: Procedure: Conventional Esthetic crown lengthening

INTERVENTIONS:
Procedure: Conventional Esthetic crown lengthening — Conventional Surgical Esthetic Crown Lengthening
  Arms: Control Group
Procedure: Computer guided Esthetic crown lengthening — Computer guided Esthetic crown lengthening
  Arms: Test Group

SUMMARY:
The objective of the present study was to evaluate the effectiveness of surgical esthetic crown lengthening using digitally assisted 3D printed surgical stents in management of excessive gingival display due to altered passive eruption.

DETAILED DESCRIPTION:
The objective of the present study was to evaluate the effectiveness of surgical esthetic crown lengthening using digitally assisted 3D printed surgical stents in management of excessive gingival display due to altered passive eruption.

Primary objectives:

Wound healing Score: the clinical features of periodontal wound healing were measured according to Hagenaars et al using the following parameters: swelling of the soft tissue , color of the gingiva, probing pocket depth, bleeding index, plaque index, clinical attachment level. These signs were assessed at 1 week, 3 months and 6 months post-operative.

Operating time: the time needed to complete each procedure was calculated in minutes by using a stopwatch from the time of the first incision till the completion of bone removal.

Secondary objectives:

Patient satisfaction: was assessed using visual analogue scale at 24 hours, 7 days and 14 days post operatively. (Zero is for minimum pain and ten is for maximum pain).

Gingival margin stability: The position of gingival margin in relation to a reference point was evaluated immediately after surgery, 3 months and 6 months healing period .

ELIGIBILITY:
Inclusion Criteria:

1. Males and females within age range of 20-40 years.
2. Systemic (medically) free individuals.
3. Excessive gingival display in the esthetic zone (more than 3mm of gingival display at full smiling)
4. Patients with good oral hygiene.

Exclusion Criteria:

1. Smokers (15)
2. Teeth with compromised periodontium.
3. Pregnant and lactating females.
4. The vulnerable group: patients with mental or physical disabilities.
5. Patients with parafunctional habits.
6. Medications that affect periodontal wound healing.
7. Periodontal surgery in the esthetic zone in the past 6 months.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Wound Healing | Change in soft tissue features from 1 week to 6 months post operative
  the clinical features of periodontal wound healing were measured according to Hagenaars et al using the following parameters: color of the gingiva (C) (a score of 0-2) 0=no redness, 1=moderate redness, 2=pronounced redness
Operating time | During surgery
  the time needed to complete each procedure from the first incision till the completion of bone removal

SECONDARY OUTCOMES:
Patient satisfaction | 1 day - 1 week - 2 weeks post operative
  will be assessed using numerical visual analogue scale (scale of zero - no pain to ten- maximum pain)
Gingival margin stability | Baseline - 3 months post operative - 6 months post operative
  The position of gingival margin in reference to an index is measured from the incisal edge to the free gingival margin

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt